CLINICAL TRIAL: NCT00994864
Title: Preoperative Chemosensitivity Testing as Predictor of Treatment Benefit in Adjuvant Stage III Colon Cancer: PePiTA Trial
Brief Title: Preoperative Chemosensitivity Testing to Predict Treatment Benefit in Adjuvant Stage III Colon Cancer
Acronym: PePiTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEPITA 001; EudraCT number: 2009-011445-13
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adjuvant FOLFOX (1 pre-operative cycle) (Other): One cycle of preoperative standard FOLFOX chemotherapy followed by eleven cycles post-operatively. PET/CT before and after the pre-operative chemotherapy cycle.
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: FOLFOX — One cycle of standard FOLFOX pre-operatively followed by 11 cycles of standard adjuvant FOLFOX chemotherapy.
  Other Names: FOLFOX-4 or equivalent

SUMMARY:
The primary working hypothesis is that preoperative chemo-sensitivity testing using fluorodeoxyglucose positron emission tomography (FDG-PET) performed before and after one course of FOLFOX (folinic acid, fluorouracil, oxaliplatin) can identify the patients that will least likely have a significant benefit from adjuvant FOLFOX for stage III colon cancer. The benefit will be analyzed by correlating the preoperative FDG-PET uptake changes to the disease free and overall survival.

DETAILED DESCRIPTION:
Patients with histological confirmed colon adenocarcinoma compatible with clinical stage II or III are eligible for study screening. Receipt of a signed informed consent and study inclusion should be done within 15 days after histological diagnosis. A usual workup for preoperative staging of colon cancer must be done not more than 1 month before study inclusion and include CEA assessment, positive histological sample for colon adenocarcinoma and chest and abdominal CT scan. After receipt of the written consent, the patient undergoes baseline PET/CT scan and donates blood samples for CTC and SNP analyses. Delay between baseline examinations and histological diagnosis must not exceed 21 days. The baseline examinations should be done within 1 week before beginning of the first course of FOLFOX chemotherapy. Thirteen to 15 days after chemotherapy, the PET/CT and blood sampling for CTC analysis are repeated. Standard surgery follows after 15 days but no more than 30 days from Day 1 of preoperative chemotherapy. Two frozen tissue cores are obtained during surgery and sent immediately in dry ice shipping to the central Tumour Bank (Jules Bordet Institute) or stored locally at -80°C to be sent in batches to the central tumour bank. Thereafter, the patient receives standard care, according to tumour pathological stage. In fully eligible patients, FOLFOX chemotherapy should be started not more than 45 days after surgery. In stage III patients otherwise ineligible, recommendation is to start FOLFOX chemotherapy within 45 days after surgery although such patients will not be included in the primary analysis. Treatment in case of stage II or stage IV colon cancer is left at investigator's discretion. Eleven courses of adjuvant FOLFOX are foreseen, in order to match the usual recommendation coming from the Mosaic Trial.

Follow-up procedures after completion of adjuvant treatment will follow standard European clinical recommendations for stage II and III patients. Clinical follow-up data will be obtained for all patients, including those with stage II disease, with a minimum follow-up time of three years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical/radiological evaluation compatible with stage III colon adenocarcinoma
* No prior chemotherapy
* No prior abdominal or pelvic irradiation
* WHO performance status 0 or 1
* Effective contraception during the study and the following six months
* Signed informed consent obtained prior to any study-specific screening procedures
* Tumour considered as curatively resectable (R0) based on standard preoperative evaluations
* White blood cell count ≥ 3×109/L with neutrophils ≥ 1.5×109/L, platelet count ≥ 100×109/L, haemoglobin ≥ 9 g/dL (5.6 mmol/L)
* Direct bilirubin ≤ 1.5×ULN; ASAT and ALAT ≤ 2.5×ULN; Alkaline phosphatase ≤ 2.5×ULN; Serum creatinine ≤ 1.5×ULN
* Delay between assessment of screening criteria and first PET/CT < 21 days
* Blood glucose < 150 mg/dl at the time of FDG administration. Insulin or oral anti-diabetic medication is not allowed on the days of PET/CT imaging.
* Compliance to the first chemotherapy course to be administered before surgery
* Delay between the first PET/CT imaging and the start of neoadjuvant FOLOFX < 7 days
* Second PET/CT imaging performed on D14 (range: D13-D15, with D1 as the first day of chemo administration)
* Delay between the second PET/CT and surgery < 7 days
* Stage III (ypTNM) as assessed after surgery
* CEA < 1.5 x ULN 1 month after surgery -

Exclusion Criteria:

* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to screening. Incompletely healed wounds or anticipation of the need for major surgical procedure during the course of the study
* Any suspicion of metastatic disease
* Rectal cancer located within 15 cm from the anal verge by endoscopy or under the peritoneal reflection at surgery
* Inflammatory bowel disease
* Pregnancy (absence to be confirmed by ß-hCG blood test) or breast-feeding
* History or current central nervous system disease or peripheral neuropathy
* Hypersensitivity to any of the components of study treatments
* Previous malignancy in the last five years except basal-cell carcinoma of the skin or in situ cervical carcinoma
* Clinically relevant coronary artery disease or history of myocardial infarction in the last 6 weeks or high risk of uncontrolled arrhythmia
* Medical, geographical, sociological, psychological or legal conditions that would not permit the patient to complete the study or sign informed consent
* Any significant disease which, in the investigator's opinion, would exclude the patient from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2009-11; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Examine the predictive value of PET-assessed tumour FDG uptake response after one course of preoperative chemotherapy on the outcome of adjuvant therapy, measured by 3-year DFS. | Within 3 years after completion of adjuvant chemotherapy

SECONDARY OUTCOMES:
Examine the predictive value of PET-assessed tumour FDG uptake changes after one course of preoperative chemotherapy on OS | Within 3 years after completion of adjuvant chemotherapy
Evaluate the best cut-off value for relative delta SUV in assessment of preoperative chemotherapy response by FDG-PET/CT imaging. | Within 3 years after completion of adjuvant chemotherapy
Analyze the cost-effectiveness of preoperative chemo-sensitivity testing | Within 3 years after completion of adjuvant chemotherapy
Assess the predictive value of circulating tumour cells on disease-free survival | Within 3 years after completion of adjuvant chemotherapy
Assess the predictive value of SNPs on toxicity- and drug target-related genes on DFS | Within 3 years after completion of adjuvant chemotherapy
Create a frozen tumour bank for future studies | Within 2 years from the beginning of study

CONTACTS AND LOCATIONS:
Overall Officials: Alain Hendlisz, MD, Principal Investigator — Jules Bordet Institute, Brussels, Belgium
Locations (21):
- Belgium (21):
  - Clinique St-Luc Bouge, Bouge
  - Hôpital Erasme, Brussels
  - Jules Bordet Institute, Brussels
  - CHU Brugmann, Brussels
  - IRIS Etterbeek-Ixelles, Brussels
  - Clin Université St-Luc Bruxelles, Brussels
  - HIS IZZ Bracops, Brussels
  - Grand Hôpital Charleroi, Charleroi
  - UZ Antwerp, Edegem
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHR Citadelle de Liege, Liège
  - CHU De Liège, Liège
  - Clinique St-Joseph, Liège
  - ZNA - Jan Palfijin, Merksem
  - CHU Ambroise Paré, Mons
  - CHR Namur, Namur
  - AZ Damiaan, Ostend
  - clinique St Pierre Ottignies, Ottignies
  - AZ Turnhout, Turnhout
  - Clinique Universites UCL Mont-Godinne, Yvoir

REFERENCES:
- [Derived] Hendlisz A, Golfinopoulos V, Deleporte A, Paesmans M, Mansy HE, Garcia C, Peeters M, Annemans L, Vandeputte C, Maetens M, Borbath I, Dresse D, Houbiers G, Fried M, Awada A, Piccart M, Laethem JL, Flamen P. Preoperative chemosensitivity testing as Predictor of Treatment benefit in Adjuvant stage III colon cancer (PePiTA): protocol of a prospective BGDO (Belgian Group for Digestive Oncology) multicentric study. BMC Cancer. 2013 Apr 12;13:190. doi: 10.1186/1471-2407-13-190. PMID 23587148